CLINICAL TRIAL: NCT06678412
Title: The Validity and Reliability of the Turkish Version of the Cognitive Functioning Self-Assessment Scale
Brief Title: Turkish Version of the Cognitive Functioning Self-Assessment Scale
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Okur, Assistant Professor, Kutahya Health Sciences University
Other Study IDs: KSBU 2024/11-09
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Impairment
Keywords: cognitive function; self-assessment; psychometrics
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Self-report scales used in the assessment of cognitive functions can serve as an initial screening tool for the general population, aside from specific neuropsychiatric tests, which are more costly and time-consuming. This study is designed to examine the validity and reliability of the Turkish version of the Cognitive Functioning Self-Assessment Scale (CFSS). Permission for the study has been obtained from the developer of the scale, Dr. Maria Antonietta Annunziata. The Turkish translation of the scale will be made, and approval will be obtained from the original author for the final version. Subsequently, the Turkish version of the CFSS, the Hospital Anxiety and Depression Scale, and the Cognitive Failures Questionnaire will be administered to participants. Surveys will be completed either online via Google Forms or in written form. To assess the reliability of the scale, the Turkish version of the CFSS will be re-administered to the same participants 7-14 days later.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years old

Exclusion Criteria:

* Taking antidepressants
* Having a neurological or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals over 18 years old
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Functioning Self-Assessment Scale (Turkish Vesion) | Baseline and 7-14 days after
  The "Cognitive Functioning Self-Assessment Scale" developed by Annunziata et al. in 2016, consists of 18 questions aimed at assessing cognitive function areas such as attention, memory, problem-solving, temporal-spatial orientation, and dual-task performance. Scoring is done on a 5-point Likert scale, ranging from 1 to 5. Higher scores on the scale indicate an increase in subjective cognitive complaints.
Hospital Anxiety and Depression Scale (HADS) | Baseline
  The HADS was developed by Zigmond and Snaith in 1983. The HADS consists of a total of 14 items, including 7 items for anxiety and 7 items for depression. The items are scored between 0-3 points on a 4-point Likert-type scale according to how the individual felt in the previous week. The scores that can be obtained from anxiety and depression subscales vary between 0-21. The Turkish validity and reliability study of the scale was conducted by Aydemir et al. in 1997. High scores obtained from the scale indicate increased mood disorder.
Cognitive Failures Questionnaire (CFQ) | Baseline
  The BDI is a self-report scale developed by Broadbent et al. in 1982 to assess cognitive failures that occur in daily life. Errors in perception, memory and motor functions are assessed with 25 questions. Each question is scored from 0 (never) to 4 (very often). The total score that can be obtained from the scale ranges from 0-100. Higher scores indicate an increased level of cognitive failure and worse cognitive status. The Turkish validity and reliability study of the scale was conducted by Ekici et al. in 2016.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)